CLINICAL TRIAL: NCT06964750
Title: Tele-Rehabilitation With Web-Based Exercises for Individuals With Postural Problems: A Digital Touch for Postural Disorders
Brief Title: the Effect of Web-based Exercises on Postural Deformities
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Tezel Yıldırım Şahan, Associate Proffessor, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Telerehabilitation on posture; Academician (Other: University of Health Sciences Turkiye)
Record Dates: First submitted 2025-03-19; First posted 2025-05-09 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Telerehabilitation; Posture; Lordosis; Kyphosis; Home Based Rehabilitation
Keywords: telerehabilitation; posture; lordosis; kyphosis; exercise
MeSH Terms: conditions — Lordosis; Kyphosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Individuals will be divided into two groups: home based exercise group and telerehabilitation group.
Masking Description: Participants will not know which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise (Experimental): Participants will practice for 6 weeks.
  Interventions: Behavioral: Exercise; Behavioral: home based exercise

INTERVENTIONS:
Behavioral: Exercise — Groups will practice the exercises by different method for 6 week
Behavioral: home based exercise — Participant were practice for 6 weeks home based exercises.

SUMMARY:
this study aims to investigate the effect of telerehabilitation with web-based exercises on postural deformities in individuals with postural problems. This randomized controlled study is planned to include 40 individuals. The individuals will be university students between the ages of 18-25. The students will be divided into two groups: home exercise program and telerehabilitation group. Exercises will be applied to both groups 3 times a week for 6 weeks.

DETAILED DESCRIPTION:
Objective: Recent studies have shown that the use of telerehabilitation in different areas can result in significant clinical gains. The effect of telerehabilitation on head forward posture, thoracic hyperkyphosis and lumbar hyperlordosis is not yet fully understood. Therefore, this study aims to investigate the effect of telerehabilitation with web-based exercises on postural deformities in individuals with postural problems.

Method: This randomized controlled study is planned to include 40 individuals. The individuals will be university students between the ages of 18-25. The students will be divided into two groups: home program and telerehabilitation group. Exercises will be applied to both groups 3 times a week for 6 weeks. Individuals with postural problems will be evaluated for craniovertebral, kyphosis and lordosis angles, shortness of hamstring and pectoral muscles and trunk endurance. Craniovertebral, kyphosis and lordosis angles will be evaluated with the "Clinometer + Buble" application, muscle shortness will be evaluated with muscle shortness tests, and trunk endurance will be evaluated with trunk endurance tests.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering for research,
* Be a young adult between the ages of 18 and 25,
* To be a student of SBU Gülhane Faculty of PTR,
* Body mass index less than 30 kg/m2,
* Cranioverterbral angle less than 52 degrees,

Exclusion Criteria:

* - Neck, back or lower back pain,
* Being a regular exerciser or professional/amateur athlete
* Having a three-dimensional deformity such as scoliosis,
* Having a previous operation, neurological, orthopedic or congenital problem in the spine,
* Visual and hearing loss that prevents them from performing the assessments and exercises,
* Physiotherapy within the last 6 months,

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
craniovertebral, lordosis, and kyphosis angles | After 6 weeks from the initial assessment
  craniovertebral angle (CVA), lordosis, and kyphosis angles will measure with a smartphone application before and after 6 weeks.

SECONDARY OUTCOMES:
shortness | After 6 weeks from the initial assessment
  Participants will evaluated with muscle shortness test on pectoral and hamstring muscles
Endurance | After 6 weeks from the initial assessment
  Participants will evaluated with trunk endurance tests.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science, Ankara, Kecioren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jeong GH, Lee BH. Effects of Telerehabilitation Combining Diaphragmatic Breathing Re-Education and Shoulder Stabilization Exercises on Neck Pain, Posture, and Function in Young Adult Men with Upper Crossed Syndrome: A Randomized Controlled Trial. J Clin Med. 2024 Mar 11;13(6):1612. doi: 10.3390/jcm13061612. PMID 38541838
- [Background] Mbada CE, Olaoye MI, Dada OO, Ayanniyi O, Johnson OE, Odole AC, Ishaya GP, Omole OJ, Makinde MO. Comparative Efficacy of Clinic-Based and Telerehabilitation Application of Mckenzie Therapy in Chronic Low-Back Pain. Int J Telerehabil. 2019 Jun 12;11(1):41-58. doi: 10.5195/ijt.2019.6260. eCollection 2019 Spring. PMID 31341546
- [Background] Lee Y, Jung KB. Effect of Physiotherapy to Correct Rounded Shoulder Posture in 30 Patients During the COVID-19 Pandemic in South Korea Using a Telerehabilitation Exercise Program to Improve Posture, Physical Function, and Reduced Pain, with Evaluation of Patient Satisfaction. Med Sci Monit. 2022 Dec 27;28:e938926. doi: 10.12659/MSM.938926. PMID 36573031
- [Background] Huang T, Zhang W, Yan B, Liu H, Girard O. Comparing Telerehabilitation and Home-based Exercise for Shoulder Disorders: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2024 Nov;105(11):2214-2223. doi: 10.1016/j.apmr.2024.02.723. Epub 2024 Mar 2. PMID 38432330